CLINICAL TRIAL: NCT04133480
Title: An Open-Label Exploratory Investigation of Cognitive Outcomes With Cannabidiol Oral Solution (EPIDIOLEX®; GWP42003-P)
Brief Title: Investigation of Cognitive Outcomes With Cannabidiol Oral Solution
Acronym: EPI-COG
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The decision to withdraw the study was based on pandemic-related concerns of conducting a Phase IV study requiring multiple clinic visits when medication is commercially available. The study was withdrawn before any participants were recruited.
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWEP18060
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Lennox-Gastaut Syndrome
Keywords: GWP42003-P; EPIDIOLEX®; cannabidiol; CBD; cognition
MeSH Terms: conditions — Lennox Gastaut Syndrome | interventions — Cannabidiol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- GWP42003-P (Experimental): For the first 7 days of the treatment period, participants are to take GWP42003-P at a dose of 5 milligrams per kilogram per day (mg/kg/day), administered as 2 equally divided doses (i.e., 2.5 mg/kg in the morning and 2.5 mg/kg in the evening). On Day 8, participants are to increase the dose to 10 mg/kg/day, administered as 2 equally divided doses (i.e., 5 mg/kg in the morning and 5 mg/kg in the evening). The 10 mg/kg/day dose should be maintained for the remainder of the treatment period; however, per labeling, investigators may increase the dose to a maximum of 20 mg/kg/day if clinically warranted by titrating an additional 5 mg/kg/day each week until reaching the maximum dose. GWP42003-P will be taken b.i.d. (morning and evening).
  Interventions: Drug: GWP42003-P

INTERVENTIONS:
Drug: GWP42003-P — oral solution of 100 milligrams per milliliter (mg/mL) cannabidiol (CBD)
  Other Names: Cannabidiol; CBD; Epidiolex

SUMMARY:
This study is being conducted to evaluate the effects of GWP42003-P on cognition in pediatric participants, aged 3 to 10 years, with Lennox-Gastaut Syndrome (LGS).

DETAILED DESCRIPTION:
This trial is a 30-week (4-week baseline period; 26-week treatment period) open-label exploratory investigation of the effects of GWP42003-P on cognitive abilities in participants with LGS who reside in the United States.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant is male or female aged 3-10 years.
* Participants' parent(s)/legal representative is willing and able to give informed consent for participation in the trial; where the participant possesses adequate understanding, informed assent should also be taken.
* Participant and their caregiver are willing and able (in the investigator's opinion) to comply with all trial requirements.
* Participant must have a clinical diagnosis of Lennox-Gastaut Syndrome (LGS), with onset within the last 5 years. This includes certification from the investigator of prior electroencephalogram (EEG) documenting slow spike wave (< 3 Hertz [Hz]) during the participant's history and evidence of more than 1 type of generalized seizure, including drop seizures (atonic, tonic, or tonic-clonic), for at least 6 months.
* Investigator can confirm that the addition of GWP42003-P to the participant's existing antiepileptic drug (AED) regimen is warranted.
* Participant must have at least 1 drop seizure each week during the first 28 days of the baseline period.
* A minimum level of general intellectual functioning as assessed at screening with the Peabody Picture Vocabulary Test
* Participant's parent(s)/legal representative is willing to allow the responsible authorities to be notified of participation in the trial, if mandated by local law.
* Participant's parent(s)/legal representative is willing to allow his or her primary care practitioner (if they have one) and consultant (if they have one) to be notified of participation in the trial, if the primary care practitioner/consultant is different to the investigator.

Key Exclusion Criteria:

* Participant has clinically significant unstable medical conditions other than epilepsy.
* Participant experiences > 300 total seizures within the first 28 days of the baseline period.
* Participant has any prior exposure to GWP42003-P.
* Participant has initiated felbamate within the last 12 months.
* Participant has initiated mammalian target of rapamycin (mTOR) inhibitors for epilepsy within the last 4 weeks.
* Participant is currently using or has in the past used recreational or medicinal cannabis or synthetic cannabinoid-based medications (including Sativex®) within the 3 months prior to trial entry.
* Participant has had clinically relevant symptoms or a clinically significant illness, other than epilepsy, in the 4 weeks prior to screening or Visit 2.
* Participant has laboratory values at screening or Visit 2 that are clinically significantly abnormal in the investigator's opinion.
* Participant tests positive for Δ9-tetrahydrocannabinol (THC) or cannabidiol (CBD) at screening.
* Participant has any known or suspected hypersensitivity to cannabinoids or any of the excipients of GWP42003-P.
* Participant has significantly impaired hepatic function at the screening visit, defined as any of the following:

  * Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 × upper limit of normal (ULN);
  * Serum ALT or AST > 3 × ULN and (total bilirubin [TBL] > 2 × ULN or international normalized ratio [INR] > 1.5);
  * Serum ALT or AST > 3 × ULN with the presence of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (> 5%).
* Participant has received an investigational medical product within the 3 months prior to the screening visit.
* Participant has any other significant disease or disorder, which, in the opinion of the investigator, may either put the participant at risk because of participation in the trial, may influence the result of the trial, or may affect the participant's ability to take part in the trial.
* Any abnormalities identified following a physical examination of the participant that, in the opinion of the investigator, would jeopardize the safety of the participant if he/she took part in the trial
* Participant has been previously enrolled into this trial.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to end of treatment (Day 181 [Visit 5]) in processing speed on the National Institutes of Health Toolbox Cognition Battery (NIHTCB) | Baseline; Day 181

SECONDARY OUTCOMES:
Change from Baseline to Day 91 (Visit 4) in processing speed on the NIHTCB | Baseline; Day 91
Change from Baseline to Day 91 (Visit 4) and Day 181 (end of treatment; Visit 5) in executive function and attention on the NIHTCB | Baseline; Days 91 and 181
Change from Baseline to Day 91 (Visit 4) and Day 181 (end of treatment; Visit 5) in episodic memory on the NIHTCB | Baseline; Days 91 and 181
Change from Baseline to Day 91 (Visit 4) and Day 181 (end of treatment; Visit 5) in language on the NIHTCB | Baseline; Days 91 and 181
Change from Baseline to Day 91 (Visit 4) and Day 181 (end of treatment; Visit 5) in the NIHTCB Childhood Composite Score | Baseline; Days 91 and 181
Change from Baseline to Day 91 (Visit 4) and Day 181 (end of treatment; Visit 5) in the Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2) or BRIEF, Preschool (BRIEF-P) for participants aged 5 years or younger | Baseline; Days 91 and 181
Change from Baseline to Day 91 (Visit 4) and Day 181 (end of treatment; Visit 5) in weekly seizure frequency | Baseline; Days 91 and 181
Change from Baseline to Day 91 (Visit 4) and Day 181 (end of treatment; Visit 5) in behavior using the Aberrant Behavior Checklist, Second Edition Community Forms (ABC-2-3) | Baseline; Days 91 and 181
Change from Baseline to Day 91 (Visit 4) and Day 181 (end of treatment; Visit 5) in sleep characteristics using the Children's Sleep Habits Questionnaire (CSHQ) | Baseline; Days 91 and 181
Change from Baseline to Day 181 (end of treatment; Visit 5) in quality of life using the Pediatric Quality of Life Inventory (PEDS-QL4) | Baseline; Day 181
Change from Baseline to Day 91 (Visit 4) and Day 181 (end of treatment; Visit 5) in generic health status using the EQ-5D-Y Proxy Version 1 | Baseline; Days 91 and 181
Change from Baseline to Day 91 (Visit 4) and Day 181 (end of treatment; Visit 5) in the Caregiver Global Impression of Change (CGIC) score | Baseline; Days 91 and 181
Change from Baseline to Day 91 (Visit 4) and Day 181 (end of treatment; Visit 5) in Patient-Reported Outcomes Measurement Information System (PROMIS®) - Parent Proxy Short Form Anxiety and Depression Subscales | Baseline; Days 91 and 181
Change from Baseline to Day 91 (Visit 4) and Day 181 (end of treatment; Visit 5) in Parenting Stress Index, Fourth Edition (PSI-4) | Baseline; Days 91 and 181
Change from Baseline to Day 181 (end of treatment; Visit 5) in the participant's ability to perform day-to-day tasks | Baseline; Day181
Change from Baseline to Day 91 (Visit 4) and Day 181 (end of treatment; Visit 5) in the Physician Global Impression of Change (PGIC) score | Baseline; Days 91 and 181
Number of participants with the indicated type of adverse event | up to Day 219
Number of participants with clinically significant changes in laboratory parameter values | Baseline; up to Day 191
Number of participants with clinically significant changes in physical examination findings | Baseline; up to Day 191
Number of participants with clinically significant changes in vital sign values | Baseline; up to Day 191

IPD SHARING:
Plan to Share IPD: No